CLINICAL TRIAL: NCT02668549
Title: Cross-Sectional Study to Define and Validate "Doctor/Pharmacy Shopping" as Outcomes Suggestive of Abuse and/or Addiction
Status: Completed | Type: Observational
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Collaborators: World Health Information Science Consultants, LLC (Other); IMS Health (Other)
Responsible Party: Sponsor
Other Study IDs: Observational Study 3033-8; 3033-8 (Other: Member Companies of the Opioid PMR Consortium)
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Patients with Opioid dispensings: Patients receiving two or more opioid dispensings within 18 months
  Interventions: Other: DB review for Doctor/Pharmacy Shopping Behavior
- Patients with Diuretic dispensings (neg control): Patients receiving two or more Diuretics dispensings within 18 months will serve as negative control
  Interventions: Other: DB review for Doctor/Pharmacy Shopping Behavior

INTERVENTIONS:
Other: DB review for Doctor/Pharmacy Shopping Behavior — Database review to evaluate of doctor/pharmacy shopping behaviors

SUMMARY:
The purpose of this study is to formulate definitions of doctor/pharmacy shopping and evaluate its association with abuse/addiction

DETAILED DESCRIPTION:
Based on a review of the literature, the Food and Drug Administration (FDA) concluded that more data are needed regarding the serious risks of misuse, abuse, addiction, overdose, and death associated with the long-term use of extended release/long acting (ER/LA) opioid analgesics. Thus, the FDA is requiring that ER/LA opioid analgesic drug sponsors conduct post-marketing studies to assess these risks. The four observational post-marketing requirement (PMR) studies are labeled Study #2065-1, Study #2065-2, Study #2065-3, and Study #2065-4.

The objective of PMR Study #2065-4 is to define and validate "doctor/pharmacy shopping" as outcomes suggestive of misuse, abuse and/or addiction.

Study #2065-4 consists of three sub-studies, Study 4A, Study 4B, and Study 4C. In the current study (#2065 sub-study, Study 4A), the IMS® LRx database, a longitudinal pharmacy database that captures both third-party and self-pay transactions, will be linked to the PharMetrics Plus™ database, which contains provider, facility and pharmacy claims. From these databases, patients with shopping behavior will be identified and evaluated against an algorithm for abuse/addiction that will be developed and validated in PMR Study #2065-3B. Study #2065-3B will review the literature for health information suggestive of abuse/addiction in medical charts and medical claims. Then, through iterative processes that involve experts reviewing claims profiles and medical charts, text searches of medical records using natural language processing and supervised machine learning will identify and create a compilation of codes and health information with the best specificity and sensitivity to identify patients with opioid abuse/addiction. The compilation of codes and health information will be used to develop the algorithm that Study 4A will apply to define abuse/addiction. Restricting the validation of shopping behavior to only patients with diagnoses related to abuse would ignore the population with undiagnosed abuse. By supplementing ICD-9 codes with other information available on claims (e.g., addiction treatments, emergency visits) to define abuse/addiction, the measurement bias will be decreased and the estimates of the association of shopping behavior with abuse/addiction will be more valid. Categories of doctor shopping will be derived from the population distributions of the multiple variables analyzed for opioid users. The 4 categories will range from no shopping behavior (lowest level) to extensive shopping behavior (most extreme). The specifics of how the categories will be defined will be driven by the data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Minimum of two dispensings for IR or ER/LA opioids or two or more diuretic dispensings

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years of age or older) with data in both IMS LRx and PharMetrics Plus, who also have a minimum of two dispensings for IR or ER/LA opioids or two or more diuretic dispensings. The first of these dispensings will have occurred in 2012 and an additional dispensing within 18 months after the first. Dispensings will be determined from the IMS LRx database.
Sampling Method: Non-Probability Sample
Enrollment: 164923 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Numbers and proportions of patients with shopping behavior | Retrospective review over 18 month period starting with first dispensing in 2012
Sensitivity and predictive value of different levels of shopping behavior in relation with Algorithmically Identified Abuse and Addiction (AIAA) | Retrospective review over 18 month period starting with first dispensing in 2012

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Cepeda, MD, PhD, Study Chair — Janssen Research & Development, LLC

REFERENCES:
- [Derived] Walker AM, Weatherby LB, Cepeda MS, Bradford DC. Information on doctor and pharmacy shopping for opioids adds little to the identification of presumptive opioid abuse disorders in health insurance claims data. Subst Abuse Rehabil. 2019 Aug 1;10:47-55. doi: 10.2147/SAR.S201725. eCollection 2019. PMID 31534380